CLINICAL TRIAL: NCT04103502
Title: In Vivo Kinematics for Subjects Having a MicroPort Medial Pivot or DePuy Attune Posterior Cruciate Retainign Total Knee Arthroplasty
Brief Title: In Vivo Kinematics for Subjects Having a MicroPort Medial Pivot or DePuy Attune PCR TKA
Acronym: TKA PCR
Status: Not yet recruiting | Type: Observational
Sponsor: The University of Tennessee, Knoxville (Other)
Collaborators: MicroPort Orthopedics Inc. (Industry)
Responsible Party: Principal Investigator, Richard Komistek, Fred M. Roddy Professor of Biomedical Engineering, The University of Tennessee, Knoxville
Other Study IDs: WIRB20181868
Record Dates: First submitted 2019-09-23; First posted 2019-09-25 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Total Knee Arthroplasty; Osteo Arthritis Knee; Knee Injuries; Knee Imlant
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- MicroPort Medial Pivot: Subjects will have been implanted with the MicroPort Medial Pivot TKA
  Interventions: Device: MicroPort Medial Pivot TKA
- DePuy Attune: Subjects will have been implanted with the DePuy Attune PCR TKA
  Interventions: Device: DePuy Attune PCR TKA

INTERVENTIONS:
Device: MicroPort Medial Pivot TKA — Subjects will have been implanted with the MicroPort Medial Pivot TKA
  Groups: MicroPort Medial Pivot
Device: DePuy Attune PCR TKA — Subjects will have been implanted with the DePuy Attune PCR TKA
  Groups: DePuy Attune

SUMMARY:
In vivo knee kinematics will be assessed for 20 subjects that have been implanted with either a MicroPort Medial Pivot or DePuy Attune posterior cruciate retaining (PCR) total knee arthroplasty (TKA) by Dr. Russell Nevins of Nevada Orthopedic & Spine Center [this is the location from which participants will be recruited].

DETAILED DESCRIPTION:
There will be ten subjects with the MicroPort implant and ten with the DePuy Attune implant; however, we will increase enrollment to 24 subjects (12 in each group) to ensure that researchers acquire the necessary 20 usable datasets for analysis and also to account for any subjects that may drop out of the study. All TKAs should be judged clinically successful based on the surgeon's evaluation and each patient's Forgotten Knee Score. Each subject should have a well-functioning prosthesis, be at least six months post-operative, and should have good-to-excellent post-operative passive flexion.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will have either a MicroPort Medial Pivot or DePuy Attune PCR TKA.
* Subjects must be at least six months post-operative.
* Participants must be judged clinically successful based on the surgeon's evaluation and their Forgotten Knee Score.
* Participants must be able to perform the required activities - stepping up and a deep knee bend.
* Subjects must be willing to sign the Informed Consent (IC) / HIPAA form to participate in the study

Exclusion Criteria:

* Pregnant, potentially pregnant or lactating females. To satisfy radiation protocol, each female subject will be asked if she is pregnant, or possibly could be pregnant. A pregnant person will not be allowed to participate in the study.
* Subjects without one of the two types of knee implants under investigation.
* Subjects who are unable to perform stepping up and deep knee bend.
* Subjects who are unwilling to sign Informed Consent/ HIPAA documents.
* Does not speak English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: There will be ten subjects with the MicroPort implant and ten with the DePuy Attune implant; however, we will increase enrollment to 24 subjects (12 in each group) to ensure that researchers acquire the necessary 20 usable datasets for analysis and also to account for any subjects that may drop out of the study. All TKAs should be judged clinically successful based on the surgeon's evaluation and each patient's Forgotten Knee Score. Each subject should have a well-functioning prosthesis, be at least six months post-operative, and should have good-to-excellent post-operative passive flexion
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Kinematics Translations during Deep Knee Bend Activity | at least 6 months post-operative
  Anterior Posterior (AP) translations of lateralfemoral condyles during deep knee bend
Kinematics during Deep Knee Bend Activity | at least 6 months post-operative
  Maximum weight-bearing flexion during DKB Axial Rotation (AR) during DKB
Kinematics Translations during step up activity | at least 6 months post-operative
  Anterior Posterior (AP) translations of lateralfemoral condyles during step up activity
Kinematics during step up activity | at least 6 months post-operative
  Maximum weight-bearing flexion during DKB Axial Rotation (AR) during step up activity

CONTACTS AND LOCATIONS:
Overall Officials: Richard Komistek, Ph.D., Principal Investigator — The University of Tennessee
Locations (3):
- United States (3):
  - Nevada Orthopedic & Spine Center, Las Vegas, Nevada
  - Platinum Training/MERIN, Las Vegas, Nevada
  - The University of Tennessee, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: No
Researchers would like to retain this study data in our secure database so as to continue to add relevant, current data to our digital collection to help us work with manufacturers in the future to create better implants that last longer and will not require revision surgery. Participants will be asked if their study data may remain a part of the University of Tennessee's Center for Musculoskeletal Research data collection for use in future studies in the IC. Identifiers are automatically removed from the database upon entry into the secure server. Data shared with sponsors is de-identified.